CLINICAL TRIAL: NCT02192086
Title: The Effect of Non-Invasive Goal Directed Fluid Administration on Graft Function in Kidney Transplantation
Brief Title: Goal Directed Fluid Administration for Kidney Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fluid Kidney Transplants
Record Dates: First submitted 2014-07-07; First posted 2014-07-16 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: End Stage Renal Disease
Keywords: Kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- goal directed fluid therapy (Experimental): The "treatment" group will initially be given a 1L bolus after induction over 20 minutes (first liter may be Lactated Ringers solution or Plasmalyte, subsequent fluid will be Plasmalyte) followed by maintenance infusion at a rate of 5mL/kg/hr until the graft kidney is removed from ice. After removing the organ from ice, the kidney recipient will be administered supplemental crystalloid until PVI is 10 or lower. Plasmalyte will be warmed in accordance to the departmental hypothermia protocol. A PVI of 12 or lower will be maintained until emergence of anesthesia, at which time the PVI monitor will be removed and all patients will be managed by existing standards (pain control, fluid replacement, hemodynamic goals, etc).
  a.At the time the treatment group begins receiving goal directed fluid therapy the anesthesia team is to wean any vasopressors aggressively with the goal of terminating infusion as quickly as is safe.
  Interventions: Other: goal directed fluid therapy
- Control Group (Active Comparator): Control patients will be given a constant infusion of crystalloid (first liter may be Lactated Ringers solution or Plasmalyte, subsequent fluid will be Plasmalyte) at a rate determined by the following: 70mL/kg for the duration of the surgery, 1L bolus after induction (over 20-30 minutes) followed by the remainder as a constant infusion determined by (70mL/kg * wt - 1000mL) / 160 minutes (using the local average of approximately 180 minutes of operative time).
  a.A Masimo PVI monitor will be placed on the patient on an extremity not affected by an AV fistula and recorded for evaluation, but no fluid administration decisions will be made based on it (providers will not have access to its values).
  Interventions: Other: Control Group

INTERVENTIONS:
Other: goal directed fluid therapy — The "treatment" group will initially be given a 1L bolus after induction over 20 minutes (first liter may be Lactated Ringers solution or Plasmalyte, subsequent fluid will be Plasmalyte) followed by maintenance infusion at a rate of 5mL/kg/hr until the graft kidney is removed from ice. After removing the organ from ice, the kidney recipient will be administered supplemental crystalloid until PVI is 10 or lower. Plasmalyte will be warmed in accordance to the departmental hypothermia protocol. A PVI of 12 or lower will be maintained until emergence of anesthesia, at which time the PVI monitor will be removed and all patients will be managed by existing standards (pain control, fluid replacement, hemodynamic goals, etc).
  a.At the time the treatment group begins receiving goal directed fluid therapy the anesthesia team is to wean any vasopressors aggressively with the goal of terminating infusion as quickly as is safe.
  Arms: goal directed fluid therapy
Other: Control Group — Control patients will be given a constant infusion of crystalloid (first liter may be Lactated Ringers solution or Plasmalyte, subsequent fluid will be Plasmalyte) at a rate determined by the following: 70mL/kg for the duration of the surgery, 1L bolus after induction (over 20-30 minutes) followed by the remainder as a constant infusion determined by (70mL/kg * wt - 1000mL) / 160 minutes (using the local average of approximately 180 minutes of operative time).
  a.A Masimo PVI monitor will be placed on the patient on an extremity not affected by an AV fistula and recorded for evaluation, but no fluid administration decisions will be made based on it (providers will not have access to its values).
  Arms: Control Group

SUMMARY:
The goal of the proposed study is to evaluate the efficacy of a goal-directed fluid administration algorithm on early graft function in patients undergoing kidney transplantation. Fluid administration has increasingly been scrutinized within anesthesia related literature as an area for improvement, and the imbalance present between estimated blood loss and total fluid administered for kidney transplants must be amongst the highest case categories. Considering the patients are anuric for the majority of the procedure, unguided administration of multiple liters of crystalloid appears antiquated.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease requiring dialysis
* age >18y
* normal cognitive function.

Exclusion Criteria:

* severe left ventricular dysfunction (EF<50%)
* known cardiomyopathy
* symptomatic CAD known valvular disease
* severe anemia (Hgb<7.0)
* patients with prior transplants o
* patients who suffered surgical complications as communicated by the surgical team.

We chose these exclusion criteria to prevent enrolling patients who would not tolerate aggressive hydration possible in the treatment group. The exclusion criteria may be excessively restrictive, however, given the current practice that frequently results in rapid large volume loading without a monitor of intravascular volume status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Effect of Plethysmography Directed Fluid Administration Tranplanted Kidney | 1 year
  To determine the effect of plethysmography directed fluid administration on the incidence of delayed graft function in kidney transplantation.The treatment group will recieve fluid in a well described short period around the time of anastomosis based on a fingertip adhesive monitor. By preventing hypovolemia at the time of reperfusion, we expect the transplanted kidney to demonstrate improved function in the near term.
Pleth Variability | 1 year
  Pleth Variability Index (PVI) is a validated non-invasive monitoring method used to assess intravascular volume status, and may prove superior to dosing fluids based on existing parameters (heart rate, blood pressure, anecdotal protocols).

CONTACTS AND LOCATIONS:
Overall Officials: William Hand, MD, Principal Investigator — Medical University of South Carolina; Scott T Reeves, MD, Study Chair — Medical University of South Carolina